CLINICAL TRIAL: NCT01295554
Title: Comparative Study of Non-enhanced Versus Contrast Enhanced MR Angiography in Peripheral Arterial Disease on a 3T MR Scanner.
Acronym: AngioIRMNative
Status: Completed | Type: Observational
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: LOC/10-03 - AngioIRM-Native; 2010-A00342-37 (Other: ID RCB from AFSSAPS)
Record Dates: First submitted 2011-02-11; First posted 2011-02-14 (Estimated); Last update posted 2012-02-13 (Estimated); Status verified 2012-02

CONDITIONS: Peripheral Arterial Disease
Keywords: Peripheral arterial disease, MRA
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Peripheral arterial disease: Peripheral arterial disease
  Interventions: Other: NCE MRA and CE MRA

INTERVENTIONS:
Other: NCE MRA and CE MRA — Each patient will receive on the same day:
  * NCE MRA
  * CE MRA usually performed in the clinical routine
  After each MRA examination, the CE images will be interpreted by a radiologist and the report transmitted to the prescriber within the usual delay. The radiologists in charge of this interpretation will not be involved in the evaluation of NCE images nor in the comparison between CE and NCE images.

SUMMARY:
Magnetic Resonance Angiography (MRA) of the peripheral arteries has become essential in the diagnosis and follow-up of peripheral arterial disease.

In clinical routine, the acquisition uses intravenous injection of a Gadolinium based contrast agent (gadolinium chelates).

Initially, contrast enhanced MR angiography (CE-MRA) was recommended for diabetic patients, elderly patients and\or patients with chronic renal insufficiency presenting a contraindication to CT angiography using iodized contrast agent injection.

However, the increase in nephrogenic systematic fibrosis clinical cases, which would be secondary to gadolinium chelates injection, in patients with chronic renal insufficiency has restricted the use of CE-MRA. More than 500 cases were described to date in the world.

Its occurrence is currently estimated around 4 % for patients in terminal chronic renal insufficiency and its mortality around 30 %.

According to the recommendations of AFSSAPS from August, 2007, two gadolinium contrast agents (Gadodiamide-OMNISCAN *, General Electric HealthCare and Gadopentetate Dimeglumine-MAGNEVIST *, Bayer HealthCare) are contraindicated if the glomerular filtration rate is lower than 30 ml/mn.

Non-contrast enhanced MR angiography (NCE MRA) techniques have been proposed to provide complete and non-invasive investigation of the peripheral vasculature, from the abdominal aorta to the calf, thus offering patients with chronic renal insufficiency a surrogate with no side effects.

Moreover, the use of high field (3T) MR imaging and phased array coils offers high quality images and good signal to noise ratio for peripheral vasculature analysis.

Besides, the acquisition can be repeated if required as it does not require any contrast injection.

The main objective is to evaluate the quality of the NCE images obtained for every investigated station from the abdominal aorta to the calf.

The secondary objective is to compare the diagnostic performances of NCE images with those of CE MRA.

The third objective is to estimate the contribution of automated and dedicated post-processing tools in optimizing the diagnostic quality of the images.

DETAILED DESCRIPTION:
20 patients will be recruited either by the vascular surgery or by the cardiology departments The appointment for MRA of the peripheral arteries on the Siemens 3T MR Scanner will be given as usual.

ELIGIBILITY:
Inclusion Criteria:

* Any adult patient known or clinically suspected to present a peripheral arterial disease, the assessment of which requires an MRA of the peripheral arteries.
* MRA will be prescribed by the vascular surgery or cardiology departments. The patient should be conscious and cooperative. Clear and intelligible oral and written information will be given to the patient. The patients giving written informed consent will be included in the study.

Exclusion Criteria:

* A contraindication to MRI, in particular pacemakers or implantable defibrillators, cochlear implants, neurosurgical clips, intra-orbital or brain metallic foreign bodies, endo prothesis since less than 4 weeks or osteosynthesis material since less than 6 weeks
* Contraindication to the injection of contrast agent: pregnancy, lactation, history of allergic reaction to contrast agent injection.
* Hemodynamically unstability, acute respiratory failure, a precarious condition or a need for continuous monitoring incompatible with the constraints of MR imaging.
* Age under 18 or under legal protection measure or without social coverage.
* A refusal or inability of obtaining informed consent from the patient.

Patients withdrawing their informed consent will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patient known or clinically suspected to present a peripheral arterial disease
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2011-02; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
To evaluate the quality of the NCE images obtained for every investigated station from the abdominal aorta to the calf. | 5 months
  To evaluate the quality of the NCE images obtained for every investigated station from the abdominal aorta to the calf.

SECONDARY OUTCOMES:
To compare the diagnostic performances of NCE images with those of CE MRA. | 5 months
  To compare the diagnostic performances of NCE images with those of CE MRA.
To estimate the contribution of automated and dedicated post-processing tools in optimizing the diagnostic quality of the images. | 5 months
  To estimate the contribution of automated and dedicated post-processing tools in optimizing the diagnostic quality of the images.

CONTACTS AND LOCATIONS:
Overall Officials: Yves Gandon, MD, Principal Investigator — Rennes University Hospital
Locations (1):
- Rennes University Hospital, Rennes, France, France